CLINICAL TRIAL: NCT01615419
Title: A Multi-national, Multi-center Non-interventional Study in Rheumatoid Arthritis (RA) Patients Treated With Tocilizumab
Brief Title: An Observational Study of RoActemra/Actemra (Tocilizumab) in Rheumatoid Arthritis Patients
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28259
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multi-center, observational study will evaluate the use in clinical practice and efficacy of RoActemra/Actemra (tocilizumab) in patients with rheumatoid arthritis. Eligible patients initiated on RoActemra/Actemra treatment according to the approved label will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe rheumatoid arthritis , according to the revised ACR criteria
* Patients initiated on RoActemra/Actemra treatment (in accordance with the local label) on their treating physicians decision

Exclusion Criteria:

* RoActemra/Actemra treatment more than 8 weeks prior to enrolment visit
* Previous RoActemra/Actemra treatment in a clinical trial or for compassionate use
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of investigational agent, whichever is longer) before starting treatment with RoActemra/Actemra
* History of autoimmune disease or of any joint inflammatory disease other than RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis initiating treatment with RoActemra/Actemra
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients on RoActemra/Actemra treatment at 6 months | approximately 2 years

SECONDARY OUTCOMES:
Rates of dose modifications/interruptions | approximately 2 years
Clinical/demographic patient characteristics at initiation of treatment | approximately 2 years
Efficacy: Response according to total joint count evaluation by DAS28/EULAR/SDAI/CDAI/ACR | approximately 2 years
Efficacy: Monotherapy versus combination therapy | approximately 2 years
Use of disease-modifying anti-rheumatic drugs (DMARDs) | approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Greece (5):
  - Athens
  - Larissa
  - Pátrai
  - Rhodes
  - Thessaloniki